CLINICAL TRIAL: NCT05656040
Title: A Single-and Multiple Dose Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of Subcutaneous MK-2060 in Participants With Chronic and/or End-Stage Kidney Disease
Brief Title: A Study of MK-2060 in Participants With Chronic and/or End-Stage Kidney Disease (MK-2060-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2060-011; MK-2060-011 (Other: MSD)
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: End-Stage Renal Disease; End-Stage Kidney Disease; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-2060 30 mg (Experimental): Participants received MK-2060 30 mg administered as a single subcutaneous dose on Day 1.
  Interventions: Biological: MK-2060
- Placebo (Placebo Comparator): Participants received placebo (normal saline) administered as a single subcutaneous dose on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: MK-2060 — MK-2060 lyophilized powder diluted in normal saline and administered subcutaneously
  Arms: MK-2060 30 mg
Drug: Placebo — Normal saline administered subcutaneously
  Arms: Placebo

SUMMARY:
This was intended as a three-part study of MK-2060 in participants with chronic and/or end-stage kidney disease (Parts 2 and 3 were not initiated due to reasons not related to safety). The purpose of Part 1 of the study was to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of a single subcutaneous dose of MK-2060 in stage 4 chronic kidney disease (CKD4) [Part2 was intended to evaluate multiple subcutaneous doses in CKD4 participants and Part 3 was intended to evaluate a single subcutaneous dose of MK-2060 in participants with end-stage kidney disease (ESRD)]. The primary hypothesis for Part 1 was that the true geometric mean of the area under the concentration-time curve from 0 to infinity (AUC0-inf) after a single-dose of MK-2060 in adult CKD4 participants would be at least 11300 nM*hr.

ELIGIBILITY:
Inclusion Criteria:

* At the time of screening, has stage 4 or 5 chronic kidney disease (Parts 1 and 2) or end-state kidney disease on peritoneal dialysis (Part 3).
* Has a body mass index (BMI) ≥ 18 and ≤ 45 kg/m^2.

Exclusion Criteria:

* Has a history of cancer, including adenocarcinoma, except adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix or other malignances which have been successfully treated ≥ 5 years prior to prestudy with appropriate follow-up.
* Has a history of deep vein thrombosis or pulmonary embolism, a history of vascular access thrombosis within 1 month prior to enrollment, or has a personal or family history of bleeding disorder.
* Has a history of gastrointestinal (GI) bleeding, duodenal polyps, or gastric ulcer in the last 5 years or severe hemorrhoidal bleed in the last 3 months.
* Has a history of or current frequent epistaxis within the last 3 months or active gingivitis.
* Has ongoing anticoagulant therapy or antiplatelet therapy. Aspirin is permitted.
* Has planned significant dental procedures at the time of screening or pre-dose or other planned surgical procedures within duration of participation of study.
* Is positive for hepatitis B surface antigen or human immunodeficiency virus (HIV).
* Has had major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-study visit.
* Has a history (participant recall) of receiving any human immunoglobulin preparation such as intravenous immunoglobulin (IVIG) or RhoGAM within the last year.
* Has a history (participant recall) of receiving any biological therapy (including human blood products or monoclonal antibodies; excluding erythropoietin and insulin) within the last 3 months or vaccination within the last 1 month, except the seasonal flu and pneumococcal vaccine or COVID-19 vaccine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Velocity Clinical Research, New Smyrna Beach ( Site 0003), Edgewater, Florida
  - Advanced Pharma CR, LLC ( Site 0006), Miami, Florida
  - Genesis Clinical Research, LLC ( Site 0004), Tampa, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0002), Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with stage 4 chronic kidney disease (CKD4) were recruited.
Groups:
- Placebo: Participants receive placebo (normal saline) administered as a single subcutaneous dose on Day 1.
Period: Overall Study
Arm/Group | MK-2060 30 mg | Placebo
Started | 11 | 3
Completed | 11 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-2060 30 mg | Placebo | Total
Number analyzed (Participants) | 11 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (9.4) | 59.0 (17.4) | 68.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Who Experience One or More Bleeding Related Adverse Events (AE)
Description: Bleeding related AEs will include any sign or symptom of bleeding, even if not requiring intervention by a medical/healthcare professional, as well as clinically relevant nonmajor bleeding or major bleeding.
Time Frame: Up to approximately 104 days
Population: All treated participants in Part 1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 3
Participants | 0 | 0

2. Primary Outcome: Part 2: Number of Participants Who Experience One or More Bleeding Related AEs
Description: Bleeding related AEs include any sign or symptom of bleeding, even if not requiring intervention by a medical/healthcare professional, as well as clinically relevant nonmajor bleeding or major bleeding.
Time Frame: Up to approximately 144 days
Population: Part 2 was never initiated.
Groups:
- MK-2060 30 mg: Participants receive MK-2060 30 mg administered as a single subcutaneous dose on Day 1.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Part 3: Number of Participants Who Experience One or More Bleeding Related AEs
Description: as for outcome 1
Time Frame: Up to approximately 104 days
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Part 1: Number of Participants Who Experience One or More AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to approximately 104 days
Population: All treated participants in Part 1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 3
Participants | 5 | 2

5. Primary Outcome: Part 2: Number of Participants Who Experience One or More AEs
Description: as for outcome 4
Time Frame: Up to approximately 144 days
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Part 3: Number of Participants Who Experience One or More AEs
Description: as for outcome 4
Time Frame: Up to approximately 104 days
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Part 1: Number of Participants Who Discontinue Study Treatment to an AE
Description: as for outcome 4
Time Frame: Up to approximately 104 days
Population: All treated participants in Part 1 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 3
Participants | 0 | 0

8. Primary Outcome: Part 2: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: as for outcome 4
Time Frame: Up to approximately 144 days
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Part 3: Number of Participants Who Discontinue Study Due to an AE
Description: as for outcome 4
Time Frame: Up to approximately 104 days
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Part 1: Area Under the Concentration-Time Curve From 0 to Infinity (AUC0-inf) of MK-2060
Description: Blood was collected to determine the AUC0-inf of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and 90 post-dose
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 0
hr*nM | 14300 (40.9) |

11. Primary Outcome: Part 2: AUC0-inf of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the AUC0-inf of MK-2060 in plasma.
Time Frame: Days 1, 2, 4, 8, 15, and 22: pre-dose; once daily on Days 10, 17, 26, 29, 35, 42, 49, 63, 81, 111, and 130 post-dose
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Part 3: AUC0-inf of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the AUC0-inf of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 42, 60, 90, and 120 post-dose
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Part 1: Area Under the Concentration-Time Curve From Time 0 to 168 Hours (AUC0-168) of MK-2060
Description: Blood was collected to determine the AUC0-168 of MK-2060 in plasma.
Time Frame: Pre-dose, 1, 12, 24, 48, 120, and 168 hours post-dose
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 0
hr*nM | 727 (103.3) |

14. Primary Outcome: Part 2: AUC0-168 of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the AUC0-168 of MK-2060 in plasma from 0 to 168 hours.
Time Frame: Pre-dose, 24, 72, and 168 hours post-dose
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Part 3: AUC0-168 of MK-2060
Description: as for outcome 14
Time Frame: Pre-dose, 1, 12, 24, 48, 120, and 168 hours post-dose
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of MK-2060
Description: Blood was collected at pre-specified time points to determine the Cmax of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and 90 post-dose
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 0
nM | 11.3 (38.8) |

17. Primary Outcome: Part 2: Cmax of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the Cmax of MK-2060 in plasma.
Time Frame: Days 1, 2, 4, 8, 15, and 22: pre-dose; once daily on Days 10, 17, 26, 29, 35, 42, 49, 63, 81, 111, and 130 post-dose
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Part 3: Cmax of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the Cmax of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 42, 60, 90, and 120 post-dose
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Part 1: Plasma Concentration at 168 Hours (C168) of MK-2060
Description: Blood was collected at 168 hours post-dose to determine the C168 of MK-2060 in plasma.
Time Frame: 168 hours post-dose
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 0
nM | 7.19 (79.7) |

20. Primary Outcome: Part 2: C168 of MK-2060
Description: Blood was to be collected at 168 hours post-dose to determine the C168 of MK-2060 in plasma.
Time Frame: 168 hours post-dose
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Part 3: C168 of MK-2060
Description: Blood was to be collected at 168 hours post-dose to determine the C168 of MK-2060 in plasma.
Time Frame: 168 hours post-dose
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Part 1: Time to Maximum Plasma Concentration (Tmax) of MK-2060
Description: Blood was collected at pre-specified time points to determine the Tmax of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and 90 post-dose
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Median (Full Range); unit: hours
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 0
hours | 312.82 [143.67 to 648.88] |

23. Primary Outcome: Part 2: Tmax of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the Tmax of MK-2060 in plasma.
Time Frame: Days 1, 2, 4, 8, 15, and 22: pre-dose; once daily on Days 10, 17, 26, 29, 35, 42, 49, 63, 81, 111, and 130 post-dose
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Part 3: Tmax of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the Tmax of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 42, 60, 90, and 120 post-dose
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

25. Primary Outcome: Part 1: Terminal Half Life (t1/2) of MK-2060
Description: Blood was collected at pre-specified time points to determine the terminal t1/2 of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and 90 post-dose
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 0
hours | 677 (26.3) |

26. Primary Outcome: Part 2: t1/2 of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the terminal t1/2 of MK-2060 in plasma.
Time Frame: Days 1, 2, 4, 8, 15, and 22: pre-dose; once daily on Days 10, 17, 26, 29, 35, 42, 49, 63, 81, 111, and 130 post-dose
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Part 3: t1/2 of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the terminal t1/2 of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 42, 60, 90, and 120 post-dose
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

28. Primary Outcome: Part 1: Apparent Total Clearance (CL/F) of MK-2060
Description: Blood was collected at pre-specified time points to determine the CL/F of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and 90 post-dose
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 0
Liters/hour | 0.0141 (40.9) |

29. Primary Outcome: Part 2: CL/F of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the CL/F of MK-2060 in plasma.
Time Frame: Days 1, 2, 4, 8, 15, and 22: pre-dose; once daily on Days 10, 17, 26, 29, 35, 42, 49, 63, 81, 111, and 130 post-dose
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

30. Primary Outcome: Part 3: CL/F of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the CL/F of MK-2060 in plasma.
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 42, 60, 90, and 120 post-dose
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

31. Primary Outcome: Part 1: Apparent Volume of Distribution (Vz/F) of MK-2060
Description: Blood was collected at pre-specified time points to determine the Vz/F of MK-2060 in plasma
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and 90 post-dose
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 11 | 0
Liters | 13.8 (39.6) |

32. Primary Outcome: Part 2: Vz/F of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the Vz/F of MK-2060 in plasma
Time Frame: Days 1, 2, 4, 8, 15, and 22: pre-dose; once daily on Days 10, 17, 26, 29, 35, 42, 49, 63, 81, 111, and 130 post-dose
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

33. Primary Outcome: Part 3: Vz/F of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the Vz/F of MK-2060 in plasma
Time Frame: Day 1: pre-dose, 1 and 12 hours post-dose; once daily on Days 2, 3, 6, 8, 11, 14, 21, 28, 42, 60, 90, and 120 post-dose
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Part 1: Mean Fold Change From Baseline in Activated Partial Thromboplastin Time (aPTT) of MK-2060
Description: Blood was collected at pre-specified time points to determine the aPTT of MK-2060 in plasma. Positive and negative scores indicate increases and decreases, respectively, in aPTT compared to baseline.
Time Frame: Day 1 (1 hr and 12 hrs postdose) and Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and Post Study (Day 90)
Population: All Part 1 participants treated with MK-2060 and who have data available are included.
Measure: Mean (Standard Error); unit: Mean fold change from baseline
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 9 | 3
Mean fold change from baseline
  Day 1: 1 Hour Postdose: number analyzed (Participants) | 7 | 2
  Day 1: 1 Hour Postdose | 1.047 (0.028) | 0.977 (0.037)
  Day 1: 12 Hours Postdose | 1.044 (0.03) | 0.994 (0.017)
  Day 2: number analyzed (Participants) | 7 | 2
  Day 2 | 1.05 (0.021) | 0.971 (0.02)
  Day 3 | 1.137 (0.04) | 1.032 (0.033)
  Day 6 | 1.219 (0.059) | 1.075 (0.081)
  Day 8 | 1.202 (0.059) | 1.08 (0.093)
  Day 11 | 1.157 (0.063) | 1.08 (0.084)
  Day 14 | 1.128 (0.042) | 1.102 (0.114)
  Day 21 | 1.114 (0.037) | 1.01 (0.075)
  Day 28: number analyzed (Participants) | 8 | 3
  Day 28 | 1.07 (0.048) | 1.012 (0.049)
  Day 60: number analyzed (Participants) | 8 | 3
  Day 60 | 1.101 (0.038) | 1.053 (0.115)
  Post Study (Day 90) | 1.026 (0.044) | 1.129 (0.064)

35. Secondary Outcome: Part 2: Percent Change From Baseline in aPTT of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the aPTT of MK-2060 in plasma.
Time Frame: Day 1 (1 hr and 12 hrs postdose) and Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and Post Study (Day 90)
Population: Part 2 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Part 3: Percent Change From Baseline in aPTT of MK-2060
Description: Blood was to be collected at pre-specified time points to determine the aPTT of MK-2060 in plasma.
Time Frame: Day 1 (1 hr and 12 hrs postdose) and Days 2, 3, 6, 8, 11, 14, 21, 28, 60, and Post Study (Day 90)
Population: Part 3 was never initiated.
Arm/Group | MK-2060 30 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 104 days
Description: All treated participants are included.
Arm/Group | MK-2060 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/3
Other Adverse Events (participants affected / at risk) | 5/11 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2060 30 mg (N=11) | Placebo (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2060 30 mg (N=11) | Placebo (N=3)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT05656040/Prot_SAP_000.pdf